CLINICAL TRIAL: NCT05159947
Title: Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Trial of the Efficacy and Safety of SPT-07A Injection in Patients With Acute Ischemic Stroke
Brief Title: SPT-07A Injection in Patients With Acute Ischemic Stroke (AIS): A Phase III Clinical Trial
Acronym: SPAIR-2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Suzhou Huyun New Drug Research and Development Co., Ltd (Unknown); Shanghai Canming Pharmaceutical Technology Co., Ltd (Unknown); Beijing Haijinge Pharmaceutical Technology Co., Ltd (Unknown); The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science and Technology (Unknown); Xiang Yang NO.1 People's Hospital (Unknown); Xiangyang Central Hospital (Other); Wuhan NO. 4 hospital (Unknown); The Affiliated Hospital of Xuzhou Medical University (Other); Xuzhou Central Hospital (Other); Yan'an University Xianyang hospital Co., Ltd (Unknown); Hengshui People's Hospital (Other); Inner Mongolia Baogang Hospital (Other); Daqing oilfield general hospital (Unknown); The Fourth Affiliated Hospital of Harbin Medical University (Other); The First Hospital of Jilin University (Other); Meihekou Central Hospital (Unknown); Jiangsu Taizhou People's Hospital (Other); Tianjin People's Hospital (Other); Taizhou Hospital (Other); Zhejiang Taizhou hospital (Unknown); The First Affiliated Hospital of Nanhua University (Unknown); Jining Medical University (Other); Zhongshan Hospital Xiamen University (Other); Neijiang Second People's Hospital (Unknown); Tancheng first people's Hospital (Unknown); The Affiliated Hospital of Qingdao University (Other); Taian Central Hospital (Unknown); Weihai Municipal Hospital (Other); Nanyang nanshai hospital (Unknown); Dezhou People's Hospital (Other); The First Affiliated Hospital of Nanyang Medical College (Unknown); Deyang People's Hospital (Other); Yantai Yuhuangding Hospital (Other); Qingdao Central Hospital (Other); Fukuang General Hospital of Liaoning health industry group (Unknown); Xi'an Gaoxin Hospital (Other); Affiliated Hospital of Jiaxing University (Other); Fujian Zhangzhou hospital (Unknown); The Affiliated Hospital of Inner Mongolia Medical University (Other); Daqing people's Hospital (Unknown); Hainan People's Hospital (Other); Qujing first people's Hospital (Unknown); The Third Affiliated Hospital of Qiqihar Medical College (Unknown); The First Affiliated Hospital of Hebei North University (Other); Linfen Central Hospital (Unknown); Xuancheng people's hospital (Unknown); The First Affiliated Hospital of Shihezi University Medical College (Unknown); Guangzhou Red Cross Hospital (Other); People's Hospital of Wuhan University (Unknown); Wuhan Central Hospital (Other); Jingzhou Central Hospital (Other); The Central Hospital of Huanggang (Other); Sinopharm Dongfeng General Hospital (Unknown); Changjiang Shipping General Hospital (Unknown); Yichang Central People's Hospital (Other); The Central Hospital of Enshi Tujia And Miao Autonomous Prefecture (Other); Xiangtan Central Hospital (Other)
Responsible Party: Principal Investigator, Hu Bo, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPT-07A
Record Dates: First submitted 2021-12-07; First posted 2021-12-16 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (SPT-07A injection group) (Experimental)
  Interventions: Drug: SPT-07A injection
- Control group (placebo group) (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: SPT-07A injection — 20mg (2), dissolved in 250ml of normal saline, and injected intravenously for 90±20min, twice a day, and administered for 7 days.
  Arms: Test group (SPT-07A injection group)
Other: placebo — 2 Injection simulants, dissolved in 250ml of normal saline, and injected intravenously for 90±20min, twice a day, and administered for 7 days.
  Arms: Control group (placebo group)

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel controlled clinical trial in Chinese patients with acute ischemic stroke. Objective to evaluate the efficacy and safety of SPT-07A injection compared with placebo in the treatment of patients with acute ischemic stroke.

DETAILED DESCRIPTION:
The target population of this study is patients with acute ischemic stroke within 48 hours. All potential participants must provide informed consent, and those who provide informed consent will enter the screening (- 48 ~ 0h), and the screening qualification will be evaluated according to the inclusion criteria. The eligible subjects will enter the treatment period (day 1-7) and will be randomly assigned to the experimental group (SPT-07A injection group) or the control group (placebo group).

During the treatment period, all subjects will receive SPT-07A injection or placebo by intravenous drip, twice a day for 7 consecutive days. During the treatment, all subjects need to receive basic treatment: citicoline sodium injection 0.25g, intravenous drip slowly, once a day, continuous administration for 7 days. According to the Chinese guidelines for the diagnosis and treatment of acute ischemic stroke (2018), the patients were given antihypertensive, hypoglycemic, lipid-lowering, anticoagulant or mannitol. All subjects were not allowed to receive interventional therapy (mechanical thrombectomy or stent implantation, etc.), thrombolysis (such as rtPA and urokinase), other cerebrovascular dilators (such as Butylphthalide, Flunarizine, Nicardipine and Nimodipine, etc.), other neuroprotective agents (such as Edaravone,etc., except citicoline) during the whole trial period. After the end of the treatment period (the 7th day), the subjects will enter the follow-up period (the 8th-90th day).

During the follow-up period, subjects need to be followed up twice (30th day ± 3 days, 90th day ± 7 days).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 to 85 years;
2. According to the Key points for diagnosis of various major cerebrovascular diseases in China 2019 and combined with the experience of clinicians, patients with ischemic stroke were diagnosed;
3. From "the last time that looks normal" to the beginning of drug treatment ≤ 48 hours. When the onset time of symptoms can not be accurately obtained after awakening stroke or due to aphasia, disturbance of consciousness and other reasons, the final time of normal performance of patients should be taken as the criterion.
4. First onset of ischemic stroke or prestroke with mRS of 0 or 1;
5. A National Institutes of Health Stroke Scale (NIHSS) score between 6 and 20, and a total score of upper and lower limbs ≥2 on motor deficits;
6. Capable of understanding the purpose and risk of the study and has signed, in writing, the informed consent form (ICF). If the subject is not capable of this at the time of enrollment, a legally authorized representative (LAR) will provide written informed consent in accordance with all regulations.

Exclusion Criteria:

1. Serious disturbance of consciousness (NIHSS 1a ≥2 score);
2. Based on the opinion of the Investigator, the posterior circulation symptoms like ataxia in stroke patients are caused by posterior circulation ischemia, such as brainstem or cerebellum;
3. Neuroimaging (CT/MRI) revealed intracranial hemorrhagic diseases (such as cerebral hemorrhage, epidural hematoma, subdural hematoma, subarachnoid hemorrhage, ventricular hemorrhage, traumatic cerebral hemorrhage, etc.);
4. Rapidly improving or resolving symptoms, suggesting a possible transient ischemic attack (TIA) rather than a qualifying stroke;
5. Subjects who are ready to undergo or have undergone intravenous thrombolysis, or endovascular therapy in 90 days from onset;
6. Renal insufficiency: Serum creatinine > 2.5 times the upper limit of normal value, or other known serious renal insufficiency diseases;
7. Liver function damage: ALT and AST > 2.5 times the upper limit of normal value, or other known liver diseases such as acute and chronic hepatitis, cirrhosis, etc.;
8. Poorly controlled hypertension, with systolic blood pressure (≥ 180 mmHg) and/or diastolic blood pressure ( ≥110 mmHg);
9. Subjects with heart rate < 40 beats/min and/or heart rate > 120 beats/min; 2-degree or 3-degree cardiac block without pacemaker or other malignant arrhythmia; acute myocardial infarction or interventional therapy in the past month, patients with heart failure (according to NYHA grade III-IV);
10. Patients with status epilepticus who are unable to cooperate or unwilling to cooperate due to other organic mental disorders and moderate or severe cognitive impairment;
11. Subjects with malignant tumors, serious diseases of the blood, digestive or other systems or hemophilia and the expected survival time is not more than 3 months;
12. Female subjects who are pregnant, lactating/breast-feeding, or plan to become pregnant;
13. Allergic constitution, or allergic to experimental drugs, analogous drugs or basic treatment drugs;
14. Received treatment with any other investigational drug within 30 days before Baseline, or is currently participating in another clinical study;
15. Any other reasons that, in the opinion of the investigator, make the subject unsuitable for enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1112 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-01-10 (Estimated); Study Completion 2024-01-10 (Estimated)

PRIMARY OUTCOMES:
Good outcome at 90 days | at day 90 (±7)
  proportion of subjects with a modified Rankin Scale (mRS) ≤ 1

SECONDARY OUTCOMES:
proportion of subjects with a modified Rankin Scale (mRS) ≤ 2 at day 90(±7) | at day 90(±7)
  proportion of subjects with a modified Rankin Scale (mRS) ≤ 2
National Institute of Health stroke scale (NIHSS) at day 8(+1) | at day 8(+1)
  proportion of subjects with a National Institute of Health stroke scale (NIHSS) 0-1 or mean improvement value from baseline
Barthel Index (BI) at day 90(±7) | at day 90(±7)
  proportion of subjects with a Barthel Index (BI) ≥95
modified Rankin Scale (mRS) at day 8(+1), 30(±3) and day 90(±7) | at day 8(+1), 30(±3) and day 90(±7)
  score of modified Rankin Scale (mRS)
National Institute of Health stroke scale (NIHSS) at day 8(+1), 30(±3) and day 90(±7) | at day 8(+1), 30(±3) and day 90(±7)
  score of National Institute of Health stroke scale (NIHSS)
Barthel Index (BI) at day 8(+1), 30(±3) and day 90(±7) | at day 8(+1), 30(±3) and day 90(±7)
  score of Barthel Index (BI)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Hu, Dr. or PhD., Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No